CLINICAL TRIAL: NCT04510792
Title: IMpact of hyPeRkalaemia on thErapy With Renin angiotenSin aldoSterone System Inhibitors
Acronym: IMPRESS
Status: Withdrawn | Type: Observational
Why Stopped: withdrawn
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/60
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hyperkalemia
Keywords: Hyperkalemia due to RAASi; RAASi; Hyperkalaemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
There are limited data regarding the burden of hyperkalaemia in patients attending emergency departments (ED) or who are hospitalised (excluding those already receiving dialysis). Renin-angiotensin-aldosterone system inhibitors (RAASi) are of prognostic benefit in patients with heart failure with reduced ejection fraction (HFrEF) and post myocardial infarction (MI) left ventricular systolic dysfunction (LVSD) and as such should be continued wherever possible for these indications. These drugs may contribute to elevation in serum potassium and hyperkalaemia may lead to a reduction in dose or complete withdrawal of RAASi. Yet it remains unknown how common this happens in standard clinical practice. Inappropriate discontinuation of RAASi in such patients may lead to adverse clinical outcomes. If patients have hyperkalaemia that limits the use of RAASi, they may be candidates for new potassium binders that could facilitate their continued use.

DETAILED DESCRIPTION:
Research questions:

In an adult population of patients who are hospitalised or attending the emergency department (and not receiving dialysis) with hyperkalaemia:

1. How does hyperkalaemia impact on RAASi therapy and does this vary according to the clinical indication for the drug(s)?
2. What are the demographics, co-morbidities and drug history for patients presenting with hyperkalaemia?
3. What is the frequency of subsequent hospitalisations and mortality rate in a cohort of patients presenting with hyperkalaemia at 12 months?

ELIGIBILITY:
Inclusion Criteria:

1. Patients in ED or inpatients with at least 1 blood test with a potassium level of ≥5.5 mmol/l
2. Receiving RAASi.
3. Aged 18 and above.
4. Able to provide informed consent or consent provided by consultee in those unable to consent for themselves.

Exclusion Criteria:

1. Patients already receiving dialysis prior to the episode of hyperkalaemia.
2. For patients considered for postal consent: known cognitive impairment, learning difficulties or brain injury or those who had transient cognitive impairment, delirium or required urgent deprivation of liberty form completion during inpatient stay or in the previous 12 months prior to hyperkalaemia episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients or ED attenders receiving RAASi and with an episode of hyperkalaemia (potassium ≥5.5 mmol/l)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who take RAASi for clear prognostic indications and who had changes to RAASi as a result of hyperkalaemia. | 12 months
  Proportion of hospitalised patients/ED attenders receiving RAASi for clear prognostic indication who experience RAASi dose reduction/withdrawal due to hyperkalaemia at discharge.
Proportion of patients who take RAASi without clear prognostic indications and who had changes to RAASi as a result of hyperkalaemia. | 12 months
  Proportion of hospitalised patients/ED attenders receiving RAASi without clear prognostic indication who experience RAASi dose reduction/withdrawal due to hyperkalaemia at discharge.

SECONDARY OUTCOMES:
Recurrent hyperkalaemias. | 12 months
  Number of repeated episodes of hyperkalaemia after initial episode according to laboratory reports (episodes can be as inpatient or outpatient) captured during study period.
Proportion of patients continuing of RAASi. | 3 months and 12 months
  Proportion of patients continuing of RAASi therapy after initial episodes of hyperkalaemia at 3 months and 12 months.
Hospitalisations | 12 months
  Number and causes (all cause, cardiovascular or HF) of hospitalisations at 12 months
Mortality | 12 months
  Number and causes (all cause, cardiovascular or HF) of mortality at 12 months.
Level of hyperkalaemia leading to changes to RAASi. | 12 months
  Level of hyperkalaemia at which healthcare professionals reduce dose/stop RAASi.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Kalra, Professor, Principal Investigator — Portsmouth Hospitals University NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No